CLINICAL TRIAL: NCT03497117
Title: 19F Magnetic Resonance Imaging of Ventilation in Subjects With Cystic Fibrosis Undergoing Treatment for Pulmonary Exacerbation
Brief Title: 19F MRI of Ventilation in Subjects With Cystic Fibrosis Undergoing Treatment for Pulmonary Exacerbation
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Enrollment barriers made study completion impossible
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15-0239; 2P30DK065988-11 (NIH)
Record Dates: First submitted 2018-03-29; First posted 2018-04-13 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Cystic Fibrosis
Keywords: imaging; hyperpolarized; perfluorinated; MRI; lung; multiple breath washout; lung clearance index
MeSH Terms: conditions — Cystic Fibrosis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: Participants undergoing treatment for a pulmonary exacerbation will perform multiple breath washout and undergo an MRI with inhalation of a gas contrast agent (79% perfluoropropane (PFP) mixed with 21% oxygen) at the beginning and end of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CF pulmonary exacerbation group (Other): Patients with cystic fibrosis being treated for a pulmonary exacerbation will undergo Lung Clearance Index (LCI) and an MRI with PFP.
  LCI testing will take place before the MRI. Each test will take 5-20 minutes and up to three tests will be performed with at least 5-minute rest periods between each test.
  PFP gas will be administered using a full-face mask during the MRI. Images are acquired during 12-second breath-hold after every 3rd breath. Before and after the MRI is complete, participants will perform spirometry maneuvers in a room outside of the magnet.
  Interventions: Device: Lung Clearance Index; Drug: MRI with PFP

INTERVENTIONS:
Device: Lung Clearance Index — To assess the efficiency of ventilation distribution and gas mixing by measuring the rate of clearance of an inert gas (nitrogen) from the lungs.
  Other Names: LCI
Drug: MRI with PFP — * Description: inhaled PFP, a gaseous contrast agent (79% PFP, 21% O2, pre-mixed, medical grade gas)
  * Administration: Full-face disposable ventilation mask and a standard Douglas Bag system.
  * Dosage: Two controlled breaths of contrast gas followed by a full breath and a 12-second breath-hold and scan for image acquisition.
  * Frequency: Repeated 5 times followed by an identical five cycles with room air to ensure PFP gas wash-out has occurred.
  Other Names: Perfluoropropane gas (C3F8); 19F

SUMMARY:
The purpose of this study is to use perfluorinated gas imaging to highlight regions of functional variation within the lungs of participants with cystic fibrosis (CF), and to correlate this with changes in spirometry, lung clearance index, and quality of life of CF subjects undergoing treatment for a pulmonary exacerbation.

DETAILED DESCRIPTION:
The investigators hypothesize that 19F-enhanced MRI will detect improvements in lung ventilation following the treatment of a CF pulmonary exacerbation, and changes in ventilation as well as global MRI scores will track with both spirometry and quality of life assessments. Therefore, investigators propose this pilot and feasibility study to gain preliminary data on a comparison of the changes in ventilation that occur with treatment of a pulmonary exacerbation, as well as to begin to understand the repeatability of this novel outcome measure. Through this study, the investigators aim to: 1) Compare quantitative and qualitative assessments of lung ventilation using 19F MRI imaging and traditional, global physiologic assessments (spirometry, LCI) and compare these with images obtained in an age-matched healthy control population; 2) Correlate changes in MRI scoring with subjective changes in health related outcomes as measured by the CFQ-R (Cystic Fibrosis Questionnaire - Revised); 3) Determine the ability of 19F MRI to detect changes in ventilation that occur with treatment of a CF pulmonary exacerbation; and 4) Determine the repeatability of 19F MRI assessment of ventilation in a disease population.

Participants with CF with baseline forced expiratory volume in 1 second (FEV1) of at least 40%, no contraindications to MRI, and oxygen saturation >90% on room air will be prospectively enrolled. Investigators will recruit a pre-defined cross-section of CF patients with mild, moderate, and severe lung disease, with approximately 4 subjects per group at the onset of a disease exacerbation requiring antibiotic intervention. The research team will obtain a pre-response MRI (within 3 days of initiating oral, inhaled, or IV antibiotic therapy), and a post-treatment MRI (within 3 days of terminating antibiotic treatment) to assess the responsiveness of 19F-MRI to a change in disease status. Each 19F-MRI study will be combined with assessments of spirometry, LCI (multiple breath nitrogen washout), and quality of life (CFQ-R quality of life tool).

19F-MRI will be performed by having each participant inhale a mixture of 79% perfluorinated propane (PFP) and 21% oxygen (pre-mixed) while using MRI to obtain 3D images. Subsequently, participants will be switched to room air, and cycled breathing will be continued while additional MRI images are captured to characterize gas wash-out. Safety measures, including pulse oximetry, will be monitored continuously, and spirometry will be performed before and after each MRI. Participants will also perform multiple breath washout maneuvers to obtain a lung clearance index, so this may be correlated to wash-out kinetics of the PFP.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers (<10 pack year history and no active smoking in the past year);
* Diagnosis of cystic fibrosis via standard sweat chloride/phenotypic features/genotyping
* Able to reproducibly perform lung function testing and have an FEV1 >30% of predicted at screening.
* No requirement for supplemental oxygen
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the trial.
* Participants must be willing and able to comply with scheduled visits and other trial procedures.
* Diagnosis of a pulmonary exacerbation according to Fuchs criteria (4 of the following 12 signs and symptoms) deemed to require antibiotic treatment, and must also include the change in lung function criterion:

  * Change in sputum
  * New or increased hemoptysis
  * Increased cough
  * Increased dyspnea
  * Malaise, fatigue, or lethargy
  * Temperature above 38deg C
  * Anorexia or weight loss
  * Sinus pain or tenderness
  * Change in sinus discharge
  * Change in physical examination of the chest
  * Decrease in pulmonary function by 10% or more from a previously recorded value
  * Radiographic change indicative of pulmonary infection

Exclusion Criteria:

* Under 18 years of age
* Active or former smokers with less than 1 years since quitting, or >10 pack-year smoking history
* Active asthma flare, as perceived by the study physician or unstable asthma characterized by advancement of asthma therapy in the last month or two courses of oral steroids in the past six months.
* Unable to undergo a 3.0-Tesla MRI of lungs and chest because of contraindications including

  1. Occupation (past or present) of machinist, welder, grinder
  2. Injury to the eye involving a metallic object
  3. Injury to the body by a metallic object (bullet, BB, shrapnel)
  4. Presence of a cardiac pacemaker or defibrillator
  5. Presence of aneurysm clips
  6. Presence of carotid artery vascular clamp
  7. Presence of neurostimulator
  8. Presence of insulin or infusion pump
  9. Presence of implanted drug infusion device that is not known to be MRI compatible (i.e., was placed outside of University of North Carolina Hospitals (UNCH) or is older than 10 years)
  10. Bone growth or fusion simulator
  11. Presence of cochlear, otologic or ear implant
  12. Any type of prosthesis (eye, penile, etc.)
  13. Artificial limb or joint
  14. Non-removable electrodes (on body, head or brain)
  15. Intravascular stents, filters or coils
  16. Shunt (spinal or intraventricular)
  17. Swan-Ganz catheter
  18. Any implant held in place by a magnet
  19. Transdermal delivery system (e.g. Nitro)
  20. Intrauterine device (IUD) or diaphragm
  21. Tattooed makeup (eyeliner, lips, etc.) or tattoos covering >25% of body surface area
  22. Body piercings (MUST BE REMOVED BEFORE MRI)
  23. Any metal fragments
  24. Internal pacing wires
  25. Metal or wire mesh implants
  26. Hearing aid (REMOVE BEFORE MRI) aa. Dentures (REMOVE BEFORE MRI) bb. Claustrophobia
* Unable to tolerate inhalation of the gas mixture
* Unable to adequately complete other study measures, including spirometry and multiple breath nitrogen washout
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or may interfere with the interpretation of trial results and, in the judgment of the PI, would make the participant inappropriate for enrollment.
* Pregnancy; women of childbearing potential must have a confirmed negative serum pregnancy test at screening, and a negative urine test on the day of the MRI scan, prior to the MRI scan (if serum test not performed the same day).
* Facial hair preventing a tight fit of the mask used in the study
* Allergy or intolerance due to side effects to bronchodilators

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-08-25 (Actual); Primary Completion 2019-09-13 (Actual); Study Completion 2019-09-13 (Actual)

PRIMARY OUTCOMES:
Whole lung ventilation defect volume (VDV) | 1 day
  To obtain ventilation defect volumes (VDVs), investigators will use the final wash-in image to identify all regions of interest having a signal intensity below the pre-defined threshold which indicates poor ventilation. The combined volume of all these 'ventilation defect' regions will be computed to obtain the VDV.

SECONDARY OUTCOMES:
The wash-in kinetics of PFP | 1 day
  For each participant, an exponential model will be fit to obtain a statistical estimate, T, of the rate constant that characterizes the kinetics of gas wash-in. Aggregating across all participants, the frequency distributions of T values will be characterized by tabulating estimates of the mean and standard deviation (SD). Corresponding 95% confidence intervals and the minimum, maximum, and interquartile range of T values will also be tabulated.
Ventilation defect percent (VDP) correlation with LCI | 1 day
  Changes in VDP from pre/post treatment will be correlated with changes in LCI pre- and post-exacerbation.
Ventilation defect percent (VDP) correlation with FEV1 | 1 day
  Changes in VDP from pre/post treatment will be correlated with changes in FEV1 pre- and post- exacerbation.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Goralski, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Halaweish AF, Moon RE, Foster WM, Soher BJ, McAdams HP, MacFall JR, Ainslie MD, MacIntyre NR, Charles HC. Perfluoropropane gas as a magnetic resonance lung imaging contrast agent in humans. Chest. 2013 Oct;144(4):1300-1310. doi: 10.1378/chest.12-2597. PMID 23722696
- [Background] Couch MJ, Ball IK, Li T, Fox MS, Littlefield SL, Biman B, Albert MS. Pulmonary ultrashort echo time 19F MR imaging with inhaled fluorinated gas mixtures in healthy volunteers: feasibility. Radiology. 2013 Dec;269(3):903-9. doi: 10.1148/radiol.13130609. Epub 2013 Oct 28. PMID 23985278